CLINICAL TRIAL: NCT01550497
Title: Effectiveness of Spinal Stabilization Exercises for Low Back Pain in Adolescents With Idiopathic Scoliosis
Brief Title: Spinal Stabilization Exercises for Low Back Pain in Adolescents With Idiopathic Scoliosis
Acronym: LBPAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: American Physical Therapy Association (Other); Texas Woman's University (Other)
Responsible Party: Principal Investigator, Karina Zapata, PT, DPT, PhD, physical therapist, Texas Scottish Rite Hospital for Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 092011-073
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2020-10

CONDITIONS: Adolescent Idiopathic Scoliosis; Low Back Pain
Keywords: back pain; scoliosis; home exercise program
MeSH Terms: conditions — Low Back Pain; Back Pain; Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Exercise Group (Experimental): Perform home exercises of unsupervised spinal stabilization exercises for 8 weeks
  Interventions: Other: supervised spinal stabilization exercises
- Weeky Physical Therapy Group (Experimental): weekly physical therapy of supervised spinal stabilization exercises for 8 weeks
  Interventions: Other: supervised spinal stabilization exercises

INTERVENTIONS:
Other: supervised spinal stabilization exercises — Supervised or unsupervised exercises to be done for 20 minutes at home, at least 5 times a week for the first 2 weeks and at least 3 times a week after 2 weeks. The supervised weekly physical therapy group will complete 8 weeks of weekly physical therapy. The unsupervised home exercise group will complete 8 weeks of a prescribed home exercise program.

SUMMARY:
1. Do spinal stabilization exercises demonstrate immediate and long-term effects of weight weeks of spinal stabilization exercises as measured by pain intensity and quality of life scores?
2. Does eight weeks of spinal stabilization exercises improve back muscle endurance in adolescents with Idiopathic Scoliosis (IS) with low back pain (LBP), compared to a one-time treatment (control)?

Hypotheses:

The research hypothesis for Question 1 is: Participants who receive eight weeks of spinal stabilization exercises will demonstrate significantly improved pain intensity and quality of life scores compared to participants who receive a one-time treatment after eight weeks of the intervention period and at six-month follow-up.

The research hypothesis for Question 2 is: Participants who receive eight weeks of the spinal stabilization exercises will demonstrate significantly improved back muscle endurance, compared to participants who receive a one-time treatment after eight weeks of intervention.

DETAILED DESCRIPTION:
Although idiopathic scoliosis (IS) is the most common type of scoliosis, no studies have evaluated the effectiveness of physical therapy exercises for managing low back pain (LBP) in this population. Spinal stabilization exercises are of particular importance in adolescents with IS due to possible reduced spinal stability from structural deformity. Spinal stabilization exercises have been reported to prevent recurrent episodes of LBP in the adult population. However, standardized treatment options cannot be recommended for LBP in adolescents with IS, because the investigators are not certain if spinal stabilization exercises will have the same effect on this patient population. Given the high prevalence of LBP in AIS and limited evidence of conservative interventions, researching the effectiveness of spinal stabilization exercises is warranted.

Currently, there are two common practices for managing adolescents with IS who have LBP: 1) supervised physical therapy and 2) a one-time treatment with no follow-up. No studies have examined which of these two approaches is superior. This study will provide information on optimal management of LBP in AIS. If there is no difference in outcomes between these two approaches, a one-time visit will be the optimal choice of treatment since it is more cost-effective and less burdensome for the family. If the outcomes favor the eight-week supervised physical therapy, specifically the spinal stabilization exercises, this treatment approach should be recommended for managing LBP in AIS.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 10-17),
* Idiopathic Scoliosis,
* Low Back Pain (> 2/10 on Numeric Pain Rating Scale)

Exclusion Criteria:

* other pathology of lumbar spine (like spondylotic lesion),
* current treatment (like bracing and chiropractic care),
* back pain located beyond the lumbar spine

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-03-01; Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Change in pain from initial visit | Initial visit 'day 1', After 8 weeks, After 6 months
  Numeric Pain Rating Scale

SECONDARY OUTCOMES:
Change in back muscle endurance from initial visit | Initial visit 'day 1', After 8 weeks, After 6 months
  Prone double leg raise
Change in quality of life since initial visit | Initial visit 'day 1', After 8 weeks, After 6 months
  SRS-22

CONTACTS AND LOCATIONS:
Overall Officials: Karina A Kunder, PT, DPT, Principal Investigator — Texas Scottish Rite Hospital for Children
Locations (1):
- Texas Scottish Rite Hospital for Children, Dallas, Texas, United States